CLINICAL TRIAL: NCT01969890
Title: Phase III Study on STem cElls Mobilization in Acute Myocardial Infarction
Brief Title: STem cElls Mobilization in Acute Myocardial Infarction Outcome Trial
Acronym: STEM-AMI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Upon DSMC suggestion due to a too low enrollment rate.
Sponsor: Heart Care Foundation (Other)
Collaborators: A. Manzoni Hospital (Other); Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G112
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2018-08

CONDITIONS: Anterior Acute Myocardial Infarction; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF administration (Experimental): Granulocyte Colony-Stimulating Factor (G-CSF) administration - 5 microg/kg subcutaneous every 12 hours for 6 days
  Interventions: Drug: G-CSF administration
- standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: G-CSF administration — Zarzio - 5 microg/kg bis in die for 6 days
  Other Names: Zarzio
  Arms: G-CSF administration

SUMMARY:
The purpose of this study is to demonstrate that granulocyte colony-stimulating factor (G-CSF) therapy in addition to state-of-the-art treatment (pharmacological and non pharmacological) is safe and significantly improves clinical outcome in patients with reduced left ventricular ejection fraction (LVEF) (≤45%) after successful reperfusion for large anterior acute myocardial infarction.

DETAILED DESCRIPTION:
Post infarction heart failure (HF) remains a major cause of morbidity and mortality. In the United States, more than three million patients, and 700.000 in Italy, have cardiac failure and its most common cause is ischemic heart disease. The major goal to improve post infarction LV function would be the stimulation of neovascularization and the enhancement of regeneration of cardiac myocytes within the infarcted area. Recent experimental studies suggest that bone marrow-derived progenitor cells (BMCs) or circulating endothelial progenitor cells (cEPCs) contribute to the regeneration of infarcted myocardium, to enhance neovascularization of ischemic myocardium, to prevent cardiomyocyte apoptosis, to alter scar formation by reducing the development of myocardial fibrosis and, thereby, to improve cardiac function.

G-CSF is a hematopoietic cytokine produced by monocytes, fibroblasts and endothelial cells. G-CSF is known to have multiple functions in normal, steady-state hematopoiesis. It is routinely used to mobilize CD34+ hematopoietic stem cells from the BM into peripheral blood, thus enabling their easier collection compared to BM aspirate procedure. The proven efficacy and safety of G-CSF, both in healthy donors and patients with haematological disease, along with favourable results from studies of CD34+ cell transplantation in patients with MI or ischemia, suggest that G-CSF based BMC transplantation may have an efficacy in patients with MI.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by acute anterior ST elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) or PCI-rescue with persistent occlusion of coronary artery,
* Time symptom-to-balloon (≥3 h and ≤12h or ≤24 h if symptoms persist),
* Thrombolysis in Myocardial Infarction (TIMI) flow post PCI ≥2,
* Evidence of left ventricular (LV) dysfunction (EF biplane ≤45%) ≤24 h after revascularization,
* Men and women aged ≥18 years and ≤75 years,
* Informed consent must be signed before proceeding with any study procedure.

Exclusion Criteria:

* Previous anterior MI,
* Recent MI (within 1 month),
* Known previous LV dysfunction (EF <45%),
* Patients with angiographic evidence of coronary anatomy not suitable for PCI, or needing coronary artery bypass grafting (CABG),
* Valve disease requiring surgical correction,
* History of previous cardiac surgery or PCI on LAD within 6 months,
* Previous or current documented history of leukemia, myeloproliferative or myelodysplastic disorder,
* Previous or current documented history of malignant disease,
* Haemoglobin <10 mg/dl,
* White blood cells (WBC) >25.000 mm3,
* Platelet <50.000 mm3,
* Sepsis,
* Known HIV infection,
* Immune system diseases,
* Interstitial lung disease
* Serious concomitant medical conditions (other than ischemic heart disease),
* Pregnancy and breast feeding,
* Documented alcohol and drug abuse,
* Anticipated poor compliance.
* Current participation in a clinical trial with other investigational products
* Other cell therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2013-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The composite endpoint of: - All cause death or, - recurrence of myocardial infarction (MI) or, - hospitalization due to heart failure. | two years

SECONDARY OUTCOMES:
- All cause death and cardiovascular events | two years
  The following Cardiovascular events will be assessed:
  * recurrence of MI,
  * hospitalization due to heart failure,
  * cardiovascular death,
  * coronary revascularization,
  * fatal and non fatal stroke,
  * hospitalization due to any cause,
  * cardiovascular hospitalization,
  * resuscitation and/or appropriate automated implanted cardioverter defibrillator(AICD) therapy.

OTHER OUTCOMES:
Safety endpoints - Incidence and severity of bleeding complications, - incidence of malignancy, - incidence and intensity of serious adverse events (SAEs) and adverse drug reactions (ADRs) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Felice Achilli, MD, Study Chair — Ospedale Alessandro Manzoni - Lecco; Giulio Pompilio, MD, Study Chair — Centro Cardiologico Monzino - Milano
Locations (53):
- Italy (53):
  - Ospedali Riuniti - SOD Cardiologia Ospedaliera e UTIC, Ancona, AN
  - Ospedale Generale Provinciale CG Mazzoni - Divisione di Cardiologia, Ascoli Piceno, AP
  - Ospedale San Donato - UO Cardiologia, Arezzo, AR
  - AORN Giuseppe Moscati - UO Cardiologia-UTIC, Avellino, AV
  - Humanitas Gavazzeni - UO Cardiologia, Bergamo, BG
  - Ospedale Bolognini - Divisione di Cardiologia, Seriate, BG
  - Ospedale Maggiore - UO Cardiologia, Bologna, BO
  - Ospedale Sant'Elia - Cardiologia-UTIC, Caltanissetta, CL
  - Ospedale Moriggia Pelascini - UO Cardiologia, Gravedona, CO
  - Ospedale Sant'Anna - UOC Cardiologia, San Fermo della Battaglia, CO
  - Ospedale Maggiore - UO Cardiologia e UTIC, Crema, CR
  - Istituti Ospitalieri - UO Cardiologia, Cremona, CR
  - AOU Careggi - Cardiologia Generale 1, Florence, FI
  - IRCCS San Martino Ist. Ricerca sul Cancro - UO Cardiologia, Genova, GE
  - Ospedale della Misericordia - UO Cardiologia, Grosseto, GR
  - Presidio Ospedaliero - UO Cardiologia, Sanremo, IM
  - Ospedale Alessandro Manzoni - SCD Cardiologia, Lecco, LC
  - Ospedale Campo Marte - UO Cardiologia, Lucca, LU
  - Ospedale di Circolo - UOC Cardiologia - UTIC, Desio, MB
  - Ospedale San Gerardo - UO Cardiologia UTIC, Monza, MB
  - Ospedale Bassini - UO Cardiologia e UTIC, Cinisello Balsamo, MI
  - Ospedale Civile - UTIC - Cardiologia, Legnano, MI
  - Ospedale Fatebenefratelli e Oftalmico - Cardiologia e UCC, Milan, MI
  - Ospedale Maggiore Policlinico - Divisione di Cardiologia, Milan, MI
  - Centro Cardiologico Monzino - Terapia Intensiva Cardiologica UTIC, Milan, MI
  - Ospedale San Paolo - Divisione di Cardiologia, Milan, MI
  - Ospedale San Luca - Centro Auxologico - UO Cardiologia, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia UCC, Milan, MI
  - Ospedale L. Sacco - Divisione di Cardiologia, Milan, MI
  - Ospedale Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Istituto Clinico Humanitas - UO Cardiologia Interventistica e UTIC, Rozzano, MI
  - Presidio Ospedaliero Carlo Poma - UO Cardiologia, Mantova, MN
  - Ospedale San Francesco - Cardiologia UTIC, Nuoro, NU
  - Ospedale Giovanni Paolo II - UTIC Cardiologia, Olbia, OT
  - Ospedale Civile "Guglielmo da Saliceto" - Divisione di Cardiologia, Piacenza, PC
  - Azienda Ospedaliera Padova - Clinica Cardiologica, Padua, PD
  - AOU Pisana - UO Malattie Cardiovasc. 1-Cisanello, Pisa, PI
  - Fondazione IRCCS Policlinico San Matteo - Card. con UCC-Lab. Ricerca Sperim. Card., Pavia, PV
  - Arcispedale Santa Maria Nuova - UO Degenza Cardiologica, Reggio Emilia, RE
  - AO San Giovanni Addolorata - Cardiologia 2, Roma, RM
  - Ospedale Infermi - UO Cardiologia, Rimini, RN
  - AOUS Giovanni Di Dio Ruggi D'Aragona - UOC UTIC, Salerno, SA
  - AOU San Giovanni Battista - SCDU Cardiologia 1, Torino, TO
  - AOU Ospedali Riuniti - SOC Cardiologia - Ospedale Cattinara, Trieste, TS
  - Ospedale Ca' Foncello - UOC Cardiologia, Treviso, TV
  - Ospedale di Circolo di Busto Arsizio - Divisione di Cardiologia, Busto Arsizio, VA
  - Presidio Ospedaliero di Saronno - UOC Cardiologia, Saronno, VA
  - Ospedale di Circolo Fondazione Macchi - SSD Unità di Cure Intensive Coronariche, Varese, VA
  - Ospedale dell'Angelo - UO Cardiologia, Mestre, VE
  - Ospedale Belcolle - UOC Cardiologia UTIC Emodinamica, Viterbo, VT
  - AORN Cardarelli - UO SC Cardiologia con UTIC, Napoli
  - AOU Federico II - UTIC, Napoli
  - AO Univ. Maggiore della Carità - Cardiologia 2, Novara

REFERENCES:
- [Background] Achilli F, Malafronte C, Cesana F, Maggiolini S, Mauro C, De Ferrari GM, Lenatti L, Tespili M, Pasqualini P, Gentile F, Capogrossi MC, Maggioni A, Maseri A, Pontone G, Colombo GI, Pompilio G; STEM-AMI OUTCOME Trial Investigators. Granulocyte-colony stimulating factor for large anterior ST-elevation myocardial infarction: rationale and design of the prospective randomized phase III STEM-AMI OUTCOME trial. Am Heart J. 2015 Oct;170(4):652-658.e7. doi: 10.1016/j.ahj.2015.07.005. Epub 2015 Jul 12. PMID 26386788
- [Background] Achilli F, Pontone G, Bassetti B, Squadroni L, Campodonico J, Corrada E, Facchini C, Mircoli L, Esposito G, Scarpa D, Pidello S, Righetti S, Di Gennaro F, Guglielmo M, Muscogiuri G, Baggiano A, Limido A, Lenatti L, Di Tano G, Malafronte C, Soffici F, Ceseri M, Maggiolini S, Colombo GI, Pompilio G; STEM-AMI OUTCOME CMR Sub-Study Investigators. G-CSF for Extensive STEMI. Circ Res. 2019 Jul 19;125(3):295-306. doi: 10.1161/CIRCRESAHA.118.314617. Epub 2019 May 29. PMID 31138020
- [Derived] Achilli F, Maggiolini S, Madotto F, Bassetti B, Gentile F, Maggioni AP, Colombo GI, Pompilio G; STEM-AMI OUTCOME Trial Investigators. Granulocyte colony-stimulating factor for stem cell mobilisation in acute myocardial infarction: a randomised controlled trial. Heart. 2024 Oct 28;110(22):1316-1326. doi: 10.1136/heartjnl-2024-323926. PMID 39401872